CLINICAL TRIAL: NCT03477734
Title: A Prospective, Open, Multi-Center, Controlled Study to Evaluate the Safety, Performance and Efficacy of the CardiacSense1 for Detection of Atrial Fibrillation
Brief Title: Performance and Efficacy of the CardiacSense1 for Detection of Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CardiacSense Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CL00001
Record Dates: First submitted 2018-02-20; First posted 2018-03-26 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Atrium; Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Males and females, 50 of them diagnosed with atrial fibrillation (AF), and 50 healthy participants, at least 30% of each gender in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CS1 & heart monitor - AF patients (Experimental): Males and females diagnosed with atrial fibrillation will be fitted with the CardiacSense1 and Holter heart monitor for 24-48 hours while going about daily activities, results shall be compared and analysed
  Interventions: Device: CS1 & heart monitor
- CS1 & heart monitor -Healthy volunteers (Active Comparator): Males and females not diagnosed with atrial fibrillation will be fitted with the CardiacSense1 and Holter heart monitor for 24-48 hours while going about daily activities, results shall be compared and analysed
  Interventions: Device: CS1 & heart monitor

INTERVENTIONS:
Device: CS1 & heart monitor — Daily activities while wearing the investigational device as well as the control device

SUMMARY:
A Prospective, Open, Multi-Center, Controlled Study to Evaluate the Safety, Performance and Efficacy of the CardiacSense1 for Detection of Atrial Fibrillation.

The clinical study is intended to establish the efficacy and safety of the CardiacSense1 wearable device intended to monitor and detect heart arrhythmia, specifically atrial fibrillation (A-Fib) based on a comparison to a control device, which is an off-the-shelf cleared Holter ECG device

DETAILED DESCRIPTION:
The clinical study is intended to establish the efficacy and safety of the CardiacSense1 wearable device intended to monitor and detect heart arrhythmia, specifically atrial fibrillation (A-Fib). Study design as as follows:

100 subjects, 50 (at least 30% of each gender) with A-fib and 50 without (at least 30% of each gender).

All subjects will be measured during at least 24 hours. Primary endpoint - A-Fib detection Control: Holter device will be the reference

For PPG analysis, each one hour will be considered as an event:

If A-Fib is present for more than accumulated 5 minutes in that specific hour then it shall be considered an "A-Fib hour" If A-fib was present for less than accumulated 5 minutes then it shall be considered a "Non-A-Fib hour".

For ECG analysis, each measurement of between 1-3 minutes will be considered an event.

If A-Fib is present at that specific measurement, then it shall be considered an "A-Fib event" If A-fib was not present at that specific measurement, then it shall be considered a "Non-A-Fib hour".

Sensitivity (true positive) is defined as the percentage of Holter defined "A-fib hours"/"A-Fib event" found by PPG/ECG.

The asked sensitivity is 90%. Specificity (true negative) is defined as the percentage of Holter defined "Non-A-fib hours"/"A-Fib event" found by PPG/ECG. The required specificity is 90%.

ELIGIBILITY:
Inclusion Criteria:

* Age of eighteen (18) year and above
* Diagnosed with atrial fibrilation (Permanent of persistent), or healthy participants able to and willing to sign the informed consent form For control group-no known cardiac problems

Exclusion Criteria:

* Subjects who are currently enrolled in another clinical investigation in which the intervention might compromise the safety of the subject's participation in this study.
* Subjects with low perfusion as indicated by the watch
* Women who are pregnant or breastfeeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
CardicacSense1 atrial fibrillation detection rate | 24 to 48 hours
  Comparison of the number of atrial fibrillation sessions detected by reference comparing to PPG and ECG sensors in CardiacSense device.
Safety of CardicacSense1 | 24 to 48 hours
  Incidence and severity of device related Adverse Events

SECONDARY OUTCOMES:
Usability | 24 to 48 hours
  Ease of use of the CardiacSense1 device based on user questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Havakuk, MD, PhD, Principal Investigator — Department of Cardiology, Tel Aviv Medical Center and Sackler School of Medicine, Tel Aviv University, Israel
Locations (2):
- Israel (2):
  - Rambam Medical Center, Haifa
  - Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared. Data analysis will include comparative overall data between investigational device and control device, as well as usability data